CLINICAL TRIAL: NCT03308136
Title: The Effect of Local Anesthetic Injection Depth on Procedural Pain and Discomfort During Fluoroscopically Guided Lumbar Transforaminal Epidural Injections
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 4-2017-0683
Record Dates: First submitted 2017-09-20; First posted 2017-10-12 (Actual); Last update posted 2019-01-11 (Actual); Status verified 2019-01

CONDITIONS: Lumbar Radiculopathy Due to Spinal Nerve Compression
Keywords: epidural steroid injection; procedural pain; local Anesthetic Injection
MeSH Terms: conditions — Pain, Procedural | interventions — Anesthetics, Local; Lidocaine

STUDY DESIGN:
Intervention Model Description: subcutaneous anesthesia group (group A) muscle anesthesia group (group B)
Who Masked: Participant, Investigator
Masking Description: 1. The subjects were randomly assigned to subcutaneous anesthesia group (group A) and muscle anesthesia group (group B), and the assigned results are unknown.
  2. The Outcomes Assessor is not related to the study, and does not know its contents.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- subcutaneous anesthesia group (group A) (Experimental)
  Interventions: Procedure: 1ml of local anesthetics (1% Lidocaine) were injected into the subcutaneous layer.; Drug: 1% Lidocaine
- muscle anesthesia group (group B) (Active Comparator)
  Interventions: Procedure: 1ml of a local anesthetics (1% idocaine) are first injected into the subcutaneous layer, followed by 3~4ml of local anesthetics to the muscle layer along the expected needle pathway.; Drug: 1% Lidocaine

INTERVENTIONS:
Procedure: 1ml of local anesthetics (1% Lidocaine) were injected into the subcutaneous layer. — 1) In group A, 1ml of local anesthetics (1% Lidocaine) were injected into the subcutaneous layer.
  Arms: subcutaneous anesthesia group (group A)
Procedure: 1ml of a local anesthetics (1% idocaine) are first injected into the subcutaneous layer, followed by 3~4ml of local anesthetics to the muscle layer along the expected needle pathway. — 2) In group B, 1ml of a local anesthetics (1% Lidocaine) are first injected into the subcutaneous layer, followed by 3~4ml of local anesthetics to the muscle layer along the expected needle pathway.
  Arms: muscle anesthesia group (group B)
Drug: 1% Lidocaine — 1% Lidocaine

SUMMARY:
Lumbar Transforaminal Epidural Injection is helpful for the treatment of lumbosacral radicular pain. But needle handling during the procedure may cause pain and discomfort to the patient. At the local skin anesthesia step, local anesthetics injection to the muscle layer along the needle pathway as well as the subcutaneous layer may reduce the procedural pain. In addition, it can reduce the injection site pain that may occur after the procedure.

DETAILED DESCRIPTION:
1. A planned Fluoroscopically Guided Lumbar Transforaminal Epidural Injection should be performed after receiving the informed consent of the patient.
2. This study is single-blind because it is not possible to blind the practitioner performing the injection.
3. Subjects were randomly assigned to the subcutaneous anesthesia group (group A) and the muscle anesthesia group (group B) by a random random number table, and the possibilities for belonging to any group were all the same and can not be artificially controlled by researchers.
4. After the procedure, a resident who does not know of this study records the patient's pain and discomfort. and on follow-up visits, post injection site pain is checked.
5. Because of the large difference between the skilled and unskilled patients, the procedure in this study is performed by only one skilled practitioner

ELIGIBILITY:
Inclusion Criteria:

1. Magnetic resonance imaging (MRI) and clinical manifestations of adult men and women over 20 years of age are eligible for radiculopathy due to back nerve root compression and subject to fluoroscopically guided lumbar transforaminal epidural Injection at the suspected spinal nerveroots level.

Exclusion Criteria:

1. Blood clotting disorder
2. Infection around the site
3. Contrast agent allergy
4. Uncontrolled cardiovascular, cerebrovascular, kidney disease
5. Past history of spinal surgery (ex, spinal fusion)
6. If can not block due to Non-cooperation with subjects (ex, if you can not take the stomach)
7. Patients taking narcotic analgesics

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2017-10-16 (Actual); Primary Completion 2018-02-28 (Actual); Study Completion 2018-02-28 (Actual)

PRIMARY OUTCOMES:
Procedural Pain score (NRS) | Immediately after the procedure
  Numeric Rating Scale(NRS) score : from 0 (No pain) to 10 (worst pain imaginable)

SECONDARY OUTCOMES:
At the next outpatient visit, whether the injection site pain(Yes) or not(No) | 2 weeks
  At the next outpatient visit, subjects asked about injection site pain (Yes / No) after the last injection.

CONTACTS AND LOCATIONS:
Locations (1):
- Dept. of Anesthesiology and Pain Medicine, Yonsei University College of Medicine,, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Baek IC, Choi SY, Suh J, Kim SH. The Influence of Local Anesthesia Depth on Procedural Pain During Fluoroscopically Guided Lumbar Transforaminal Epidural Injections: A Randomized Clinical Trial. Am J Phys Med Rehabil. 2019 Apr;98(4):253-257. doi: 10.1097/PHM.0000000000001032. PMID 30153126